CLINICAL TRIAL: NCT05035628
Title: Cardiopulmonary Rehabilitation in Long COVID-19 Patients With Persistent Breathlessness and Fatigue
Acronym: COVID-Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louis Bherer (Other)
Responsible Party: Sponsor-Investigator, Louis Bherer, Associate scientific director, Direction of prevention, Montreal Heart Institute, Montreal Heart Institute
Organization: Montreal Heart Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-2956
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: COVID-19 Respiratory Infection
Keywords: COVID-19; cardiorespiratory; fitness; cognition; neurovascular coupling; brain functions; physical exercise; rehabilitation; inflammatory markers; long COVID-19; cortical pulsatility
MeSH Terms: conditions — COVID-19; Motor Activity; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: parallel assignement with 2 groups (1:1)
Who Masked: Investigator, Outcomes Assessor
Masking Description: This clinical trial is a single-blinded study. Research personnel performing the outcome assessments and investigators will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiopulmonary exercise training group (Experimental): Cardiopulmonary exercise intervention will include aerobic exercise, resistance and respiratory exercises, three sessions per week for 2 months
  Interventions: Other: Cardiopulmonary exercise training
- control group (No Intervention): Control group with no intervention.

INTERVENTIONS:
Other: Cardiopulmonary exercise training — Participants will follow a 2-month exercise training program, thrice-weekly trainings. The training sessions will start with a 5-min warmup, followed by an aerobic training (20 min) after which 20-min of resistance/muscular training will take place. The program will end with respiratory exercises and cool down period (10 min). Training will be adapted to individuals' baseline capacity as measured by the baseline cardiorespiratory test.
  A certified kinesiologist will supervise trainings. Heart rate, oxygen saturation and rating of perceived exertion (Borg Scale, 6-20) will be measured during training sessions.
  Arms: Cardiopulmonary exercise training group

SUMMARY:
The objective of this project is to assess the effects of a 2-month cardiopulmonary rehabilitation program on cardiorespiratory fitness in long COVID19 patients. Quality of life, functional capacity, functional respiratory capacity, inflammatory profile, coagulation markers, cognitive functions and brain O2 saturation will also be assessed before and after the exercise rehabilitation program.

DETAILED DESCRIPTION:
Some symptoms such as breathlessness and fatigue appear to persist for several months after COVID-19 infection in about 50% of cases. Stress, anxiety, neurological and cognitive disorders have also been reported in the long-term side effects associated with the disease. Cardiopulmonary rehabilitation programs are recognized as an essential component of the management of people with chronic respiratory disease. These programs are based on exercise training with aerobic exercises, muscle strengthening, breathing exercises. Beyond the benefit on morbi-mortality, a marked improvement in symptoms, fitness and quality of life is observed in chronic respiratory diseases. Several hospital departments, research teams and scientific organizations as the WHO recommend the use of rehabilitation programs for COVID-19 patients.

The main objective is to assess the effects of a 2-month cardiopulmonary rehabilitation program on cardiorespiratory fitness in long COVID19 patients. Secondary objectives include: to characterize baseline and intervention-related changes in quality of life, functional capacity, functional respiratory capacity, inflammatory profile, coagulation markers, cognitive functions, neurovascular coupling and cortical pulsatility.

All participants will have signed a written consent form before taking part in the study.

40 patients who have had COVID-19 with persistent breathlessness and fatigue symptoms after at least 3 months after the diagnosis will be randomly assigned to one of the 2 following study arms : 1/ cardiopulmonary exercise training program; 2/ control group.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 80
* Individuals infected by the SARS-COV2 virus, with positive PCR diagnosis
* Still having breathlessness and fatigue at least 3 months after the diagnosis of COVID-19 or patients presenting an increase of 1 point (compared to before infection) on the Modified Medical Research Council scale.
* Able to perform a maximal cardiopulmonary stress test and exercise training program in accordance with current guidelines on cardiopulmonary rehabilitation.
* Able to read, understand and sign the information and consent form.

Exclusion Criteria:

* pulmonary embolism diagnosed by scintigraphy
* Absolute and relative contraindication to exercise stress test and / or exercise training
* Recent cardiovascular events (cardiac decompensation or angioplasty or cardiac surgery, less than 1 month; valvular disease requiring surgical correction, active myopericarditis, severe ventricular arrhythmias not stabilized under treatment).
* Kidney failure requiring dialysis
* heart failure (NYHA III or IV)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness | Baseline and post-intervention at 2 months
  Maximum incremental cardiopulmonary exercise test (VO2 max (ml.kg.min)

SECONDARY OUTCOMES:
Change in 6-min walking test performance | Baseline and post-intervention at 2 months
  maximum distance performed in 6 minutes (distance, m)
Change in Functional mobility | Baseline and post-intervention at 2 months
  Timed up and Go test (s).
Change in Lower limb muscles strength | Baseline and post-intervention at 2 months
  Timed Sit-to-Stand test (s).
Change in Quality-of-life | Baseline and post-intervention at 2 months
  36-Item Short Form Health Survey (Scale ranges from 0-100, with a higher score indicating a better health status).
Change in Anxiety | Baseline and post-intervention at 2 months
  State-Trait Anxiety Inventory questionnaire (Score ranges from 20-80, with a higher score indicating higher anxiety).
Change in Anxiety | Baseline and post-intervention at 2 months
  Perceived Stress Scale questionnaire (Score ranges from 0-4, with 0 no stress,1 mild stress, 3 moderate stress and 4 severe).
Change in Sleep quality | Baseline and post-intervention at 2 months
  Pittsburgh Sleep Quality Index questionnaire (Score ranges from 0-21, with a higher score indicating worse sleep quality). severe).
Change in functional respiratory capacity | Baseline and post-intervention at 2 months
  forced expiratory volume in 1 second (L.)
Change in general cognitive functioning | Baseline and post-intervention at 2 months
  Montreal Cognitive Assessment (0-30 score, with a higher score indicating a better cognitive functioning).
Change in processing speed | Baseline and post-intervention at 2 months
  Validated remote version of neuropsychological tests (Z-score)
Change in executive functions | Baseline and post-intervention at 2 months
  Validated remote version of neuropsychological tests (Z-score)
Change in episodic memory | Baseline and post-intervention at 2 months
  Validated remote version of neuropsychological tests (Z-score)
Change in inflammatory profile | Baseline and post-intervention at 2 months
  C-reactive protein (mg/L/L)
Change in oxidative stress | Baseline and post-intervention at 2 months
  serum levels of uric acid (mg/dL), albumin (g/L)
Change in markers of coagulation | Baseline and post-intervention at 2 months
  fibrinogen (g/L)
Change in neurovascular coupling | Baseline and post-intervention at 2 months
  Changes in brain activity evoked by a N-back task and walking relative to baseline will be assessed by t-statistics maps, computed from variations of [HbO] and [HbR] measured by NIRS at the prefrontal cortex.
Change in cerebral pulsatility - cortical frontal region | Baseline and post-intervention at 2 months
  Pulsatility will be measured as the normalized difference of relative near-infrared light intensity changes between systole and diastole, using NIRS in the prefrontal cortical region.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bherer, PhD, Principal Investigator — Montreal Heart Institute; Jacques Malo, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Preventive medicine and physical activity centre (centre EPIC), Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gaudreau-Majeau F, Gagnon C, Djedaa SC, Berube B, Malo J, Iglesies-Grau J, Gayda M, Bherer L, Besnier F. Cardiopulmonary rehabilitation's influence on cognitive functions, psychological state, and sleep quality in long COVID-19 patients: A randomized controlled trial. Neuropsychol Rehabil. 2025 Mar;35(2):345-361. doi: 10.1080/09602011.2024.2338613. Epub 2024 Apr 12. PMID 38607276
- [Result] Besnier F, Malo J, Mohammadi H, Clavet S, Klai C, Martin N, Berube B, Lecchino C, Iglesies-Grau J, Vincent T, Gagnon C, Gaudreau-Majeau F, Juneau M, Simard F, L'Allier P, Nigam A, Gayda M, Bherer L. Effects of Cardiopulmonary Rehabilitation on Cardiorespiratory Fitness and Clinical Symptom Burden in Long COVID: Results From the COVID-Rehab Randomized Controlled Trial. Am J Phys Med Rehabil. 2025 Feb 1;104(2):163-171. doi: 10.1097/PHM.0000000000002559. Epub 2024 Jun 24. PMID 38917451
- [Derived] Besnier F, Berube B, Malo J, Gagnon C, Gregoire CA, Juneau M, Simard F, L'Allier P, Nigam A, Iglesies-Grau J, Vincent T, Talamonti D, Dupuy EG, Mohammadi H, Gayda M, Bherer L. Cardiopulmonary Rehabilitation in Long-COVID-19 Patients with Persistent Breathlessness and Fatigue: The COVID-Rehab Study. Int J Environ Res Public Health. 2022 Mar 31;19(7):4133. doi: 10.3390/ijerph19074133. PMID 35409815